CLINICAL TRIAL: NCT07115888
Title: Reliability and Validity Assessment of the Health-Related Quality of Life Scale Developed for Active Older Adults
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Muhammed Furkan Oruç, Physiotherapist, Marmara University
Other Study IDs: 09.2024.1584
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Active Aging Individuals Aged 65 and Over
Keywords: Active Aging; Active Older Adults; Health Related Quality of Life; Reliability; Validity; Scale Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active elderly individuals aged 65 and over: Active elderly people aged 65 and over, who have the ability to see, hear and see, and who do not go to a health center for any ongoing treatment.

SUMMARY:
INTRODUCTION You are invited to take part in this academic study because you are 65 years or older and live independently in the community.

Before participating, please read the following information carefully to understand the study's procedures. After reading, if you agree to join, you will be asked to complete some questionnaires and simple mobility tests.

BACKGROUND Programs that promote health, physical activity, social interaction, and mental stimulation are becoming more important for older adults. However, there is no clear way to measure their effectiveness.

Researchers from McGill, Exeter, Erasmus, and UT Health San Antonio universities are working together to better understand active aging. In earlier studies, over 200 people were interviewed to learn how older adults perceive active living. This study now aims to examine the physical and psychological functions associated with active living.

PURPOSE OF THE STUDY This project aims to test the reliability of the HRQL-OPAL scale and assess the level of physical and psychological function related to active aging.

STUDY PROCEDURES This research is conducted under the Department of Physiotherapy and Rehabilitation, Marmara University.

If you agree to participate:

You will first complete questionnaires (approx. 20 minutes).

Then, you will perform mobility tests (approx. 20 minutes) such as walking and changing positions. A small sensor will be placed on your shoe to measure your steps and movements.

You will not be asked to do anything unsafe or difficult, like jumping or standing on one leg.

If you agree, you may be asked to complete the HRQL-OPAL scale again two weeks later.

DURATION Total time for the first session is about 40 minutes. A second session, if agreed, will take about 20 minutes after two weeks.

BENEFITS You may not receive direct personal benefit, but the results may help improve scientific knowledge and support better ways to measure quality of life in older adults.

RISKS There are no known risks. Some questions may be sensitive, but you do not have to answer any that make you uncomfortable. All tests are widely used and supervised by trained professionals.

VOLUNTARY PARTICIPATION AND WITHDRAWAL Your participation is voluntary. You may withdraw at any time without providing a reason and without any impact on your medical care.

CONFIDENTIALITY All collected data will be coded and stored securely without using your name. Only the research team will access this information.

Results may be shared in scientific reports, but your identity will remain confidential. Data will be stored for seven years by the lead researcher.

ETHICAL REVIEW This study has been reviewed and approved by the Ethics Committee of Marmara University Faculty of Medicine.

STUDY TITLE "Reliability and Validity Study of the Health-Related Quality of Life Scale Developed for Active Older Adults"

NUMBER OF PARTICIPANTS At least 92 participants who meet the criteria are required for the study.

PARTICIPANT STATEMENT I, the undersigned, confirm that I have received detailed information about this study from Physiotherapist Muhammed Furkan ORUÇ, and I have been invited to participate as a volunteer.

I understand that all personal information will remain confidential, and the study will not affect my medical care. I am aware that I can withdraw at any time.

If any health problems occur during the study, I can contact Fzt. Muhammed Furkan ORUÇ at 0534 421 52 94 or reach the institution at Küçük Çamlıca Mah. Çilehane Yolu Cad. No:51, 34696, Üsküdar/İstanbul, Prof. Dr. Fahrettin Kerim-Nilüfer Gökay Nursing Home Elderly Care and Rehabilitation Center.

I voluntarily agree to participate in this research and will receive a signed copy of this form.

DETAILED DESCRIPTION:
INTRODUCTION

As an individual aged 65 or over who is living independently in the community, you are invited to participate in this academic study.

Before participating in this study, we ask you to read the information in this form to understand the proposed procedures. The following information explains the background, objectives, procedures, benefits, and risks of this study. Please take time to read, understand, and carefully review this information. After reading the information, you will be asked a few questions about the study. If you understand the study well and agree to participate, you will be asked to complete some questionnaires and perform a few mobility tests.

BACKGROUND

Community programs that promote health, physical activity, socialization, and mental stimulation are gaining increasing importance for older adults. These programs support activities that elderly individuals consider important for active aging. However, there is currently no definitive way to measure the outcomes of these programs.

Researchers from McGill University, the University of Exeter, Erasmus University, and UT Health San Antonio have collaborated to understand how older adults maintain an active lifestyle. In these studies, more than 200 individuals were interviewed, and their perceptions of living actively were identified. The current study aims to understand the physical and psychological abilities and emotions associated with active living.

PURPOSE OF THE STUDY

This project aims to test the reliability of the HRQL-OPAL scale and measure the extent of physical and psychological function associated with how active a person is.

DESCRIPTION OF STUDY PROCEDURES

This research is conducted under the auspices of the Department of Physiotherapy and Rehabilitation at Marmara University Faculty of Health Sciences. Assessments of your physical and psychological health will be carried out at your place of residence or, if more convenient, in a specialized mobility laboratory. If you agree to participate, you will first be asked to complete some questionnaires, which will take approximately 20 minutes.

After completing the questionnaires, you will be asked to perform a simple mobility test, which will also take around 20 minutes. These tests include walking and transitioning from one position to another. While walking, a small sensor will be attached to your shoe. This sensor will count your steps and assess how well your foot moves while walking. You will not be asked to perform any test that you or the accompanying staff member thinks you are unable or should not perform - for example, jumping or standing on one leg.

If you agree, you will be asked to complete the HRQL-OPAL scale a second time, 2 weeks later.

DURATION OF THE STUDY

Completing the questionnaires will take about 20 minutes, and the mobility tests will take about 20 minutes. This will be done only once. If you agree to complete the HRQL-OPAL scale a second time, it will be conducted two weeks later.

BENEFITS OF THE STUDY

You may or may not receive personal benefits from participating in this research project. However, we hope that the results will contribute to the advancement of scientific knowledge in this area and help identify better ways to measure what matters most to older adults.

RISKS OF THE STUDY

There are no known risks associated with participating in this study. Some people may feel uncomfortable answering health-related questions, but you are not obligated to answer any question you do not wish to. The physical tests are commonly used for mobility assessment, and trained research assistants will assist you to ensure your safety during these tests.

VOLUNTARY PARTICIPATION AND RIGHT TO WITHDRAW

Your participation in this research project is entirely voluntary.

CONFIDENTIALITY

All information collected will be coded and stored without using your name. Only the research team will have access to the records.

All information collected in this study will be kept confidential and will not be shared with anyone outside the study except as required by law. Reports, publications, or presentations resulting from this study will maintain your anonymity.

During your participation, the principal investigator and the research team will collect and record only the information necessary to achieve the scientific objectives of the study. The data will be stored for 7 years after the final publication by the principal investigator. The data may be published or shared at scientific meetings; however, your identity will not be disclosed from this information.

ETHICAL OVERSIGHT OF THE STUDY

This study has been reviewed by the Ethics Committee of Marmara University Faculty of Medicine, which is responsible for the ongoing ethical oversight of the study.

STUDY TITLE

"Reliability and Validity Study of the Health-Related Quality of Life Scale Developed for Active Older Adults"

NUMBER OF PARTICIPANTS

At least 92 participants who meet the eligibility criteria are required for the completion of the study.

PARTICIPANT'S STATEMENT

I have been informed by Physiotherapist Muhammed Furkan ORUÇ that a medical research study will be conducted at the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Marmara University, and I have been provided with the above information regarding this research. Following this information, I have been invited to participate as a "participant" in this study.

I believe that the confidentiality of my personal information, which must remain private between me and my physician, will be respected and handled with great care during this study. I have been assured that my personal information will be protected with due diligence during the use of research results for educational and scientific purposes.

I am aware that I can withdraw from the study at any time for any reason. However, I understand it would be appropriate to inform the researchers beforehand to avoid causing any inconvenience. I also acknowledge that I may be removed from the study by the researcher to avoid any harm to my medical condition. I will not be held financially responsible for any expenses related to the study, nor will I receive any payment. I have been assured that any medical intervention required due to direct or indirect consequences of the study will be provided, and I will not incur any financial burden for these interventions.

In case of any health issue during the study, I know I can contact Physiotherapist Muhammed Furkan ORUÇ at 0534 421 52 94 or reach the institution at Küçük Çamlıca Mah. Çilehane Yolu Cad. No:51, 34696, Üsküdar/İstanbul, Prof. Dr. Fahrettin Kerim-Nilüfer Gökay Nursing Home Elderly Care and Rehabilitation Center. I understand that I am not obligated to participate in this study, and I have not been subjected to any coercion. I know that if I choose not to participate, it will not negatively affect my medical care or relationship with my physician.

I fully understand all the explanations provided to me. After taking adequate time to consider independently, I have decided to participate in the aforementioned research project as a "participant" (subject). I accept this invitation with great satisfaction and willingness. A copy of this signed consent form will be provided to me.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering,
* Being 65 years of age or older,
* Living independently in the community,
* Being able to walk outdoors with or without a companion and with or without an assistive device,
* Being able to see well with or without a visual aid,
* Being able to hear well with or without a hearing aid,
* Being approved for post-examination tests by Prof. Dr. Yaşar SERTBAŞ.

Exclusion Criteria:

* Participants who: • Have a medical condition requiring ongoing hospitalization in a healthcare facility (e.g., malignant tumor, kidney or liver failure);
* Are under 65 years of age;
* Are unable to live independently in the community;
* Are unable to see, hear, or walk properly, even with a device;
* Are deemed unsuitable for post-examination testing by Prof. Dr. Yaşar SERTBAŞ; • Have severe cognitive impairment;

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals who reside in Istanbul, are over 65 years of age, are actively aging, and agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life - Older Persons of Active Living (HRQL-OPAL) | Day 1 and Day 15
  The main finding of the study is the 17-item Health Related Quality of Life - Older Persons (HRQL-OPAL) measurement tool, which was developed in 2024 by Mayo et al. as a result of a multinational study based on self-report. The response options in this tool have linear characteristics, and the total score obtained from each item-assessed on a 4-point ordinal scale-reflects the overall scale score. The scale score ranges from 0 to 51, with higher scores indicating better health-related quality of life and active living.

SECONDARY OUTCOMES:
Short Form-36 Health Survey (SF-36) | Day 1
  The Short Form-36 Health Survey (SF-36) was developed in 1992 as part of the Medical Outcomes Study, a multi-year and multi-center project aimed at explaining differences in patient outcomes. The SF-36 is a self-reported instrument that assesses overall health from both physical and mental perspectives. It consists of 36 items across 8 subscales: physical functioning, social functioning, physical role limitations, emotional role limitations, pain, general health, vitality, and mental health. The scale ranges from 0 to 100, with higher scores indicating better health status.
EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) | Day 1
  As a general quality of life scale based on self-report and available in multiple languages including Turkish, the EuroQol-5 Dimension-5 Level Questionnaire (EQ-5D-5L) was introduced in 2009 by the EuroQol Group. It was developed as a five-level version to improve the sensitivity and reduce the ceiling effect of the previously created EQ-5D-3L Questionnaire by the same group. The EQ-5D-5L consists of two parts. The first part is an index that describes health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension includes five ordered response levels. To calculate the index score, participants are asked to select the most appropriate statement for each of the five dimensions. The resulting five-digit number is converted into a value between 0 (representing death) and 1 (representing perfect health) using value sets developed by the EuroQol Group. The second part of the questionnaire is a standard visual analogue sc
Lower Extremity Functional Scale (LEFS) | Day 1
  The Lower Extremity Functional Scale (LEFS), developed in 1999 by Binkley et al., is a self-reported measure designed to identify and assess the functional status of patients with lower extremity dysfunctions. The scale consists of 20 items, each with five possible response options arranged in order. The total score ranges from 0 to 80, with higher scores indicating better functional status.
Apathy Evaluation Scale (AES) | Day 1
  The Apathy Evaluation Scale (AES) was developed in 1991 by Marin et al. This scale is designed to measure the level of apathy by assessing individuals' interest in daily activities, the pleasure they derive from these activities, and their general lack of motivation. The scale has three different versions, all containing the same items: the Clinician Version (AES-C), the Informant Version (AES-I), and the Self-Report Version (AES-S). Participants are asked to respond based on their experiences over the past four weeks. The scale consists of 18 items, each rated on a four-point Likert scale. Each item is scored from 1 (not at all) to 4 (very much), resulting in a total score ranging from 18 to 72. Items 6, 10, and 11 are reverse scored, and higher total scores indicate greater levels of apathy.
Hand Grip Strength Test | Day 1
  The Grip Strength Test is a key tool used to assess hand muscle function by measuring the maximum force generated by the forearm muscles. It is well established that grip strength declines with aging, which in turn leads to a decrease in individuals' quality of life. This test is considered a reliable indicator of many age-related health conditions and is recognized as a marker of overall muscle strength.
  In our study, the Takei brand TKK 5401 model hand dynamometer (Grip-D, Takei Scientific Instruments Co. Ltd., Tokyo, Japan) was used for the Grip Strength Test. The device displays the strength of the left and right forearm flexor muscles on a three-digit digital LCD screen in kgf units. Measurements were taken while the participant was standing, with the test arm extended at a 30° angle from the body, without bending the elbow or touching the torso. The highest value obtained was recorded, and the sum of the highest values from both hands was considered the total test score.
Sit-Rise Test (SRT) | Day 1
  The Sit-to-Stand Test (SRT) is a test developed to assess individuals' flexibility, muscle strength, physical fitness, and balance skills. Various studies have reported that this test predicts all-cause mortality. The test measures the number of supports individuals use when sitting down and standing up from the floor, without shoes, on a flat, non-slippery surface, and assigns a score accordingly. Each unsupported sit-to-stand skill is scored 5 points; the maximum total score is 10, indicating good physical fitness. One point is deducted from the total score for each point of support used (hand, forearm, knee, lateral leg, hand on knee), and 0.5 points are deducted from the total score for each loss of balance observed. No time is held during the test.
2-Minute Walk Test (2MWT) | Day 1
  The 2-Minute Walk Test (2MWT) is a shorter version of the 6-Minute Walk Test (6MWT), which is frequently used in the literature as a measure of functional capacity. This test is conducted on a track of at least 30 meters, with start and end points marked by cones. Participants walk at their normal pace for 2 minutes, and the distance covered in this time is recorded in meters. This measurement provides information about an individual's functional capacity. Longer distances are considered indicators of better functional capacity. In our study, the Heel2Toe sensor (Mate et al., 2019), which was placed on the sides of the participants' shoes and provided data collection, was used to accurately measure walking quality and collect data.
Mini Balance Evaluation Systems Test (Mini-BESTest) | Day 1
  The Mini-Balance Evaluation Systems Test (Mini-BESTest) is a scale used to assess posture and balance. It is used to explain balance disorders, fall risk, and their possible causes. Its short assessment time and lack of equipment make it easy to use. The test takes 10-15 minutes to administer. The test consists of 14 items under four headings (Anti-stimulating Postural Regulation, Reactive Postural Control, Sensory Orientation, and Dynamic Gait). Each item is scored on a three-point scale (0, 1, or 2), with a maximum total score of 28. Higher scores indicate better balance and a lower risk of falling.
Tragus Posture Test (TWT) | Day 1
  The Tragus Posture Test (TWT) was developed to objectively assess spinal mobility. In this test, the subject stands with their heels and hips against a wall to prevent rotation, and their knees extended. The subject is asked to tuck their chin in. In this position, the distance between the wall and the tragus prominence of the right ear is measured with a tape measure. Greater distances indicate poorer upper cervical posture.
Fullerton Advanced Balance Scale (FAB-T) | Day 1
  The Fullerton Advanced Balance Scale (FAB-T) is a performance-based scale that comprehensively assesses static and dynamic balance in different sensory environments. It was developed to assess the multiple dimensions that constitute balance in highly functional, independently functioning, active elderly individuals. The scale, which includes 10 individual test items, is evaluated on a 5-point scale (0-4), with a maximum score of 40. Higher scores indicate better balance ability and a lower risk of future falls. There are publications indicating that an elderly person scoring 25 or below on the test can be considered with greater than 70% confidence to be at high risk of falling and requiring urgent intervention. Administration takes approximately 10-15 minutes.
Counter Movement Jump Test (CMJ) | Day 1
  The Countermovement Jump Test (CMJ) is a test developed to assess an individual's explosive lower extremity strength. This test assesses an individual's ability to jump off the ground. The participant first stands with their feet shoulder-width apart, bends their knees, and performs a squat. Then, from this position, they attempt to jump as high as possible. Force platforms can also be used in this test, and the data obtained after the participant jumps is evaluated. Because arm swinging enhances performance, care should be taken to determine whether the arms are free or stationary during the test.
  In this study, the participant was asked to perform the Countermovement Jump (CMJ) on a non-slip mat, facing a wall, with their feet shoulder-width apart. Measurements were taken three times, and the highest value achieved was recorded as the test score in centimeters.
Symbol Digit Modalities Test (SDMT) | Day 1
  The Symbol Number Modalities Test (SDMT) was developed by Aaron Smith in 1982 to assess cognitive capacity. This test measures visual-spatial scanning, attention-concentration, and information processing speed. The test includes a kit that allows for verbal and/or written assessments. This kit contains a key that matches nine numbers and symbols. Next to the key are divided blocks of randomly arranged symbols. After the first 10 trials, the participant is asked to say the numbers corresponding to the symbols on the key as quickly as possible within 90 seconds and/or mark them on the kit. At the end of the test, the total number of correct answers is calculated, and the maximum possible score is 110. The test typically takes 5 minutes to complete, and higher scores indicate better cognitive capacity.
Raven's Standard Progressive Matrices Test (RSPMT) | Day 1
  The Raven Standard Progressive Matrices Test (RSPMT) is a scale developed by John Carlyle Raven in 1936. This test was designed to assess the general cognitive capacities of people from different cultures and languages, measuring abstract reasoning. It assesses cognitive skills such as recognition, discrimination, and analogy. For this reason, it is also known as a general intelligence test. The RSPMT is more practical than other tests because it is shorter and less affected by socioeconomic factors, sensory, and motor abilities. The test consists of five sections (A, B, C, D, and E), each with 12 patterns or designs of increasing difficulty, and a total of 60 multiple-choice questions. The first two sections (A and B) have 6 options, while the last three sections (C, D, and E) have 8 options. There is no time limit for administering the test. Scoring is based on the number of correct answers, with a maximum score of 60.

CONTACTS AND LOCATIONS:
Overall Officials: Eren Timurtaş, Assoc. Prof. Dr., Study Director — Marmara University
Locations (1):
- Marmara University Health Sciences Institute, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I have obligations regarding the confidentiality of participant data.